CLINICAL TRIAL: NCT03312725
Title: Mid-term Data Collection of the Treatment of Intracranial Aneurysms With the WEB™ Aneurysm Embolization System: a Monocentric Post-market Observational Study
Brief Title: Mid-term Data Collection of the Treatment of Intracranial Aneurysms With the WEB™ Aneurysm Embolization System
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Medical Therapy Solutions (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Other Study IDs: MTS-01
Record Dates: First submitted 2017-10-03; First posted 2017-10-18 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2017-10

CONDITIONS: Ruptured and Unruptured Intracranial Aneurysms
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ruptured or unruptured intracranial aneurysms.
  Interventions: Device: WEB aneurysm embolization system

INTERVENTIONS:
Device: WEB aneurysm embolization system — The WEB aneurysm embolization system is a class III device and consists of an implantable embolization device attached to a delivery device. The WEB is a mesh composed of single layers of braided nitinol tubes with platinum cores. The braids are held together by proximal and distal platinum/iridium radiopaque markers.

SUMMARY:
Flow disruption is a new endovascular approach for treatment of both ruptured and unruptured intracranial aneurysms, which involves placement of an endosaccular device (WEB) which modifies the blood flow at the level of the neck and induces intraaneurysmal thrombosis. The WEB was designed to treat wide-neck bifurcation aneurysms. This observational study will collect data about the routine practice in one center of using the WEB in ruptured and unruptured intracranial aneurysms. The primary objective is to evaluate its efficacy by assessing the anatomic outcome during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 80 years old.
* Patient must sign and date the informed consent form <72hrs post-procedure and prior to data registration. If patient is not able to give informed consent for himself/herself, a legally authorized representative must give informed consent on his/her behalf.
* Patient has a ruptured (Hunt and Hess grades 1, 2 or 3) or unruptured intracranial aneurysm requiring endovascular treatment.
* Aneurysm with dome-to-neck ratio ≥ 1.

Exclusion Criteria:

* Aneurysm size unfavourable for WEB implantation (aneurysm width > 10 mm or aneurysm width < 3mm).
* Patient with Hunt and Hess grades 4 or 5.
* Known to be, or suspected of being unable to comply with the study protocol (e.g. no permanent address, known to be non-compliant or presenting an unstable psychiatric history).
* Parent vessel occlusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ruptured or unruptured intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Determination of anatomic outcome: grade of occlusion of the aneurysm assessed by MRA | at 6 months follow-up
  WEB Occlusion Scale:
  WOS A: complete occlusion WOS B: complete occlusion with opacification of the proximal recess WOS C: residual neck filling WOS D: residual aneurysm filling
Determination of anatomic outcome: grade of occlusion of the aneurysm assessed by MRA | at 24 months follow-up
  WEB Occlusion Scale:
  WOS A: complete occlusion WOS B: complete occlusion with opacification of the proximal recess WOS C: residual neck filling WOS D: residual aneurysm filling

SECONDARY OUTCOMES:
Determination of procedural complications (Adverse events) during the operation | During index-procedure
  Procedural complications: aneurysm rupture, dissection, thromboembolic events (symptomatic and non-symptomatic), device protrusion through the neck of the aneurysm inside the parent artery, detachment problem, device stuck in microcatheter, bleeding.
Recording the use of additional devices during treatment to occlude the aneurysm | During index-procedure
  Possible additional devices are stent, coils, flow diverter
Determination of the occurrence of post-procedural symptomatic thromboembolic events | up to 24 months follow-up
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 6 to 8 weeks follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Determination of the technical success of the device defined as device deployment in the target aneurysm as intended by the investigator with complete apposition against the aneurysm wall. | During index-procedure
Determination of 30 day mortality | up to 30 days
Determination of overall mortality | up to 24 months
Recording of intracranial haemorrhage during follow-up | up to 24 months
Need for repeat treatment during follow-up | up to 24 months
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 6 months follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 24 months follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Defreyne, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium